CLINICAL TRIAL: NCT06145984
Title: Understanding Mechanisms of Prevention of Depression: a Mechanistic Cross-over Trial of Mindfulness vs. Fantasizing to Reduce Perseverative Cognition Underlying Vulnerability for Depression
Brief Title: Mechanisms of Change of Positive Interventions in Reducing Vulnerability for Depression
Acronym: MINDCOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019/537
Record Dates: First submitted 2023-10-09; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Depression in Remission
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness first intervention, Fantasizing second intervention (Other): Diary measures of thought patterns (experience sampling method [ESM]), behavioural measures (using the Sustained Attention to Response Task [SART]), actigraphy, (neuro)physiological measures (impedance cardiography [ICG], electrocardiography [ECG] and electroencephalogram [EEG]) and measures of depressive mood (self-report questionnaires) will be performed during the week before (pre-) the interventions and the week during (peri-) performance of the interventions. In-between pre-and peri-intervention measures, there is a one month wash-out period. In this arm mindfulness will be the first performed intervention, fantasizing the second performed intervention. The order of the interventions will be counterbalanced across participants.
  Interventions: Behavioral: Mindfulness; Behavioral: Positive Fantasizing
- Fantasizing first intervention, Mindfulness second intervention (Other): Diary measures of thought patterns (experience sampling method [ESM]), behavioural measures (using the Sustained Attention to Response Task [SART]), actigraphy, (neuro)physiological measures (impedance cardiography [ICG], electrocardiography [ECG] and electroencephalogram [EEG]) and measures of depressive mood (self-report questionnaires) will be performed during the week before (pre-) the interventions and the week during (peri-) performance of the interventions. In-between pre-and peri-intervention measures, there is a one month wash-out period. In this arm fantasizing will be the first performed intervention, mindfulness the second performed intervention. The order of the interventions will be counterbalanced across participants.
  Interventions: Behavioral: Mindfulness; Behavioral: Positive Fantasizing

INTERVENTIONS:
Behavioral: Mindfulness — Participants receive a two-hour professional training to get familiar with the basic techniques of mindfulness. The training is given by a mindfulness professional and consists of psycho-education, instructions for mindfulness and guided practice. It focuses mainly on attending to stimuli such as breathing, external sounds or bodily sensations and becoming aware of where one's attention is. After the professional training, participants receive instructions about the audio application with which participants continue performing short exercises using the learned technique every day guided by an application on their smartphone customized for this research. Specifically, participants perform one short exercise (10 min) per day for in total six days. The exercises that are being performed are: attention to breathing part 1, attention to breathing part 2, attention to sounds, attention to bodily sensations, attention to thoughts, attention to emotions and feelings.
Behavioral: Positive Fantasizing — In a two-hour training session by a professional trainer, participants get familiar with the positive fantasizing technique. Participants receive psycho-education about the role of dysfunctional beliefs. The positive fantasizing technique starts with identifying dysfunctional "beliefs and schema" and subsequently fantasize about a positive "fantasy belief". Participants are guided by the professional using imagery and experiencing thoughts and feelings that would be elicited when using their fantasy belief as if in an ideal world. After using imagery techniques, participants are asked, with help of the professional, to reflect on their experience during the fantasizing exercise and to think of how they could implement this fantasy belief more in their daily life, by adapting their fantasy belief into a more practical belief. After the training, participants are asked to perform one exercise per day using the fantasizing technique using a mobile application for six days in total.

SUMMARY:
The purpose of this study is to understand the effects of mindfulness and fantasizing in reducing perseverative cognition underlying vulnerability for depression.

DETAILED DESCRIPTION:
A cross-over design will be used comparing measures before and during both a mindfulness- and a positive fantasizing intervention period in individuals who remitted from two major depressive episodes (i.e. remitted Major Depressive Disorder (rMDD) patients) and a never-depressed control group. After checking for eligibility of the participants, participants will fill-out several questionnaires about their personal characteristics, experiences and expectations. These questionnaires will be used to study individual characteristics that could serve as treatment markers predicting the effectivity of interventions. Furthermore, diary measures of thought patterns (experience sampling method [ESM]), behavioural measures (using the Sustained Attention to Response Task [SART]), actigraphy, (neuro)physiological measures (impedance cardiography [ICG], electrocardiography [ECG] and electroencephalogram [EEG]) and measures of depressive mood (self-report questionnaires) will be performed during the week before (pre-) the interventions and the week during (peri-) performance of the interventions. In-between pre-and peri-intervention measures, there is a one month wash-out period. The order of the interventions will be counterbalanced across participants. Pre- and peri-intervention measures will be compared to study intervention effects in remitted MDD patients, remitted MDD patients vs. healthy controls and in relation with individual characteristics

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, all participants must meet all the following criteria:

* Participants should be between 18 and 60 years old. Participants should not exceed 60 years of age in order to minimize aging-related decline in information processing;
* Participants should display normal intelligence (IQ>85, as assessed with the Dutch Adult Reading Test and/or having finished an education on at least vocational level) in order to assure sufficient task comprehension.

Participants in the remitted Major Depressive Disorder group should meet the following criteria to make sure that participants are at high risk of depressive relapse and currently show no clinically relevant severity of depressive symptoms:

* Remitted participants should have experienced at least two depressive episodes, according to criteria defined by the Diagnostic Statistical Manual, version 5 (DSM-5), experienced in past ten years;
* Remitted participants should score 21 or lower on the Inventory of Depressive Symptomatology (IDS-SR30), indicative of the absence of clinically relevant depressive symptoms.

Exclusion Criteria:

Furthermore, individuals who meet any of the following criteria will be excluded from participation in this study:

* Fulfilling criteria for any current DSM-5 diagnosis as objectified with the Structured Clinical Interview for DSM-5 (SCID-5);
* Daily use of anti-depressive medication, benzodiazepines, methylphenidate, beta blockers or other medication potentially influencing electrocardiogram currently or in the last four weeks;
* Recent engagement (defined as in their last episode, or as one year prior to inclusion in case the last episode was more than a year before inclusion) in preventive cognitive therapy including the positive fantasizing technique and/or have recent experiences (defined as daily practice in the past two years for at least two weeks) with mindfulness, meditation, or mindful yoga. This criterion prevents underestimation of true effects of mindfulness and/or positive fantasizing and maximizes treatment effects;
* Participation in another clinical intervention study at the moment of inclusion in the study to prevent overlapping intervention effects.

Individuals for the Never-Depressed control group who additionally meet any of the following criteria will be excluded from participation of this study:

* Presence of symptoms of depression according to the IDS-SR30 (score > 13), to make sure participants are not currently experiencing clinically relevant depressive symptoms;
* Any life-time psychopathology of any disorder as objectified with the SCID-5.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Perseverative Cognition measured with daily Experience Sampling Methods | 7 days, 10 times per day
  Daily fluctuations in self-reported perseverative cognition using Experience Sampling Methods. The main outcome measure to assess perseverative cognition using Experience Sampling Measurement is the item asking whether participants are currently ruminating. An increase in rumination scores would indicate an increase in perseverative cognition.
Physiological correlates of perseverative cognition using heart rate measured with electrocardiogram. | 24 hours
  Physiological correlates of perseverative cognition measured as heart rate, measured with electrocardiogram.
Physiological correlates of perseverative cognition using heart rate variability measured with electrocardiogram. | 24 hours
  Physiological correlates of perseverative cognition measure das heart rate variability measured with electrocardiogram
Neurophysiological correlates of perseverative cognition using electroencephalogram during performance of the Sustained Attention to Response Task. | 40 minutes task performance while measuring electroencephalogram
  Electrophysiological correlates of perseverative cognition measured using electroencephalogram (EEG) during performance of a Sustained Attention to Response Task. The Sustained Attention to Response Task is a Go/No-Go Task interrupted by thought probes asking participants about the content and characteristics of their current thoughts. While performing the task, EEG is measured. To measure the neurophysiological correlates of perseverative cognition, EEG voltage when participants reported perseverative cognition on the Sustained Attention to Response Task will be examined and and compared with the EEG voltage when participants did not report perseverative cognition.
Apathy Evaluation Scale | At baseline before the start of the measurement weeks
  Self-report questionnaire measuring apathy levels (higher score reflects higher apathy levels) examined as an individual characteristic that could be a potential individual treatment marker in predicting the effectivity of the interventions.
Bermond-Vorst Alexithymia Questionnaire | At baseline before the start of the measurement weeks
  Self-report questionnaire measuring alexithymia levels (higher score reflects higher alexithymia levels) examined as an individual characteristic that could be a potential individual treatment marker in predicting the effectivity of the interventions.
Leiden Index of Depression Sensitivity | At baseline before the start of the measurement weeks
  Self-report questionnaire measuring cognitive reactivity to sadness (higher score reflects higher cognitive reactivity) examined as an individual characteristic that could be a potential individual treatment marker in predicting the effectivity of the interventions.
Childhood Trauma Questionnaire-Short Form | At baseline before the start of the measurement weeks
  Self-report questionnaire measuring childhood trauma (higher score reflects higher childhood trauma levels) as an individual characteristic that are potential individual treatment markers in predicting the effectivity of the interventions.
Dysfunctional Attitude Scale | At baseline before the start of the measurement weeks
  Self-report questionnaire measuring dysfunctional attitudes (higher score reflects higher dysfunctional attitudes) examined as an individual characteristic that could be a potential individual treatment marker in predicting the effectivity of the interventions.
Neuroticism-Extraversion-Openness Five-Factor Inventory | At baseline before the start of the measurement weeks
  Self-report questionnaire measuring personality characteristics Neuroticism, Extraversion and Openness. The scores on these personality characteristics will be used as individual characteristics that are potential individual treatment markers in predicting the effectivity of the interventions.

SECONDARY OUTCOMES:
Inventory of Depressive Symptomatology | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring depressive symptoms (higher scores reflect higher depressive symptoms)
Perseverative Thinking Questionnaire | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring perseverative thinking (higher scores reflect higher levels of perseverative thinking)
Responses on Positive Affect Scale | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring ruminative and dampening thoughts in response to positive affect (higher scores reflect higher rumination levels).
Emotion Regulation Questionnaire | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring the emotion regulation strategies suppression and reappraisal (higher scores reflect using a particular strategy more).
Five Facet Mindfulness Questionnaire | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring five facets of mindfulness: non-reactivity to inner experience, observing, acting with awareness, describing and non-judging of experience.
Leuven Adaptation of the Rumination on Sadness Scale | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring ruminative thinking on sadness (higher scores reflect higher levels of ruminative thinking).
Positive and Negative Affect Schedule | Measured on day 7 at the end of each measurement week.
  Self-report questionnaire measuring positive and negative affect (higher scores reflect higher levels of positive or negative affect).
Sleep as measured with Actigraphy | 7 days
  Actigraphy is used as a measure of sleep-wake cycles, using the MotionWare 8. This is a device that can measure activity counts and sleep using accelerometer data interpreted by software algorithms. Actigraphy will be used to assess sleep efficacy during the measurement weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-José van Tol, professor, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Besten ME, van Vugt M, Riese H, Bockting CLH, Ostafin BD, Aleman A, van Tol MJ. Understanding mechanisms of depression prevention: study protocol of a randomized cross-over trial to investigate mechanisms of mindfulness and positive fantasizing as intervention techniques for reducing perseverative cognition in remitted depressed individuals. BMC Psychiatry. 2024 Feb 19;24(1):141. doi: 10.1186/s12888-024-05592-8. PMID 38373948